CLINICAL TRIAL: NCT01735526
Title: Changes in Lung Diffusing Capacity for Nitric Oxide and Carbon Monoxide After Allogeneic Versus Autologous Hematopoietic Stem-cell Transplantation
Brief Title: Lung Diffusing Capacity for Nitric Oxide and Carbon Monoxide After Hematopoietic Stem-cell Transplantation
Acronym: DLNO/DLCO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: 33/2012
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Lung Disease
Keywords: Allogeneic and autologous; hematopoietic stem-cell transplantation; Lung diffusing capacity; for nitric oxide; carbon monoxide; Lung tissue density; microvascular damage
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Early after allogeneic hematopoietic stem-cell transplantation (allo-HSCT), reductions of absolute lung volume and diffusing capacity for carbon monoxide (DLCO) are frequently detected even in the absence of overt idiopathic pneumonia syndrome (IPS). It can be hypothesized that these changes might be due to an occult intersitial lung disease associated with infections, acute Graft-versus-Host Disease (aGvHD), myeloablative conditioning regimens or any combination of these. To test this hypothesis, we will simultaneously measure the lung diffusing capacity for nitric oxide (DLNO) and DLCO and estimate the changes of membrane diffusing capacity (DM) and pulmonary capillary volume (Vc) by the DLNO/DLCO ratio. As we hypothesize that GHVD should be intuitively absent amongst autologous HSCT (auto-HSCT) recipients, we will compare the changes in DLNO/DLCO ratio showed by the latter group with those of subjects undergoing allo-HSCT.

DETAILED DESCRIPTION:
In allogeneic hematopoietic stem-cell transplantation (allo-HSCT) recipients, early reductions of absolute lung volume and diffusing capacity for carbon monoxide (DLCO) are frequently detected even in the absence of overt idiopathic pneumonia syndrome (IPS)[PMID: 22221781]. Two months after allo-HSCT, we have recently shown an increase in lung tissue density determined by quantitative CT scan [PMID: 22898044]. It can be hypothesized that these parenchymal changes might be due to an occult intersitial lung disease associated with infections, acute Graft-versus-Host Disease (aGvHD), myeloablative conditioning regimens or any combination of these [PMID: 21531955]. To test this hypothesis, we will simultaneously measure the lung diffusing capacity for nitric oxide (DLNO) and DLCO. Assuming, for clinical purposes, that the reaction rate of NO with blood hemoglobin is infinite so that DLNO = DMNO = DMCO*alpha (alpha = NO/CO diffusivity ratio), as to partition the effect of HSCT on membrane diffusing capacity (DM) and pulmonary capillary volume (Vc) we will use the DLNO/DLCO ratio [PMID:16478855]. As we hypothesize that GHVD should be intuitively absent amongst autologous HSCT (auto-HSCT) recipients, we will compare the changes in DLNO/DLCO ratio showed by the latter group with those of subjects undergoing allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* baseline spirometry, lung volumes, and DLCO of the subjects included in the analysis must be within the predicted normal range
* all patients must be in stable clinical conditions at the time of study

Exclusion Criteria:

* a history of bronchial asthma, chronic obstructive pulmonary disease, or other significant respiratory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing allogeneic and autologous HSCT for hematological malignancies.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in DLNO/DLCO ratio after allo- versus autologous HSCT | Before and 2-6 months after HSCT

SECONDARY OUTCOMES:
Changes in lung tissue density after allo- versus autologous HSCT | Before and 2-6 months after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barisione, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy

REFERENCES:
- [Background] Bacigalupo A, Chien J, Barisione G, Pavletic S. Late pulmonary complications after allogeneic hematopoietic stem cell transplantation: diagnosis, monitoring, prevention, and treatment. Semin Hematol. 2012 Jan;49(1):15-24. doi: 10.1053/j.seminhematol.2011.10.005. PMID 22221781
- [Background] Barisione G, Pompilio PP, Bacigalupo A, Brusasco C, Cioe A, Dellaca RL, Lamparelli T, Garlaschi A, Pellegrino R, Brusasco V. Airway distensibility with lung inflation after allogeneic haematopoietic stem-cell transplantation. Respir Physiol Neurobiol. 2012 Oct 15;184(1):80-5. doi: 10.1016/j.resp.2012.07.021. Epub 2012 Aug 8. PMID 22898044
- [Background] Panoskaltsis-Mortari A, Griese M, Madtes DK, Belperio JA, Haddad IY, Folz RJ, Cooke KR; American Thoracic Society Committee on Idiopathic Pneumonia Syndrome. An official American Thoracic Society research statement: noninfectious lung injury after hematopoietic stem cell transplantation: idiopathic pneumonia syndrome. Am J Respir Crit Care Med. 2011 May 1;183(9):1262-79. doi: 10.1164/rccm.2007-413ST. PMID 21531955
- [Background] van der Lee I, Zanen P, Grutters JC, Snijder RJ, van den Bosch JMM. Diffusing capacity for nitric oxide and carbon monoxide in patients with diffuse parenchymal lung disease and pulmonary arterial hypertension. Chest. 2006 Feb;129(2):378-383. doi: 10.1378/chest.129.2.378. PMID 16478855
- [Derived] Barisione G, Bacigalupo A, Brusasco C, Scanarotti C, Penco S, Bassi AM, Lamparelli T, Garlaschi A, Pellegrino R, Brusasco V. Mechanisms for reduced pulmonary diffusing capacity in haematopoietic stem-cell transplantation recipients. Respir Physiol Neurobiol. 2014 Apr 1;194:54-61. doi: 10.1016/j.resp.2014.01.018. Epub 2014 Feb 1. PMID 24495442